CLINICAL TRIAL: NCT03561207
Title: 3D-PREDICT REGISTRY: 3D Prediction of Patient-specific Response Using Ex Vivo Interrogation of Live Cells From Tumors
Brief Title: 3D Prediction of Patient-Specific Response
Acronym: 3D-PREDICT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KIYATEC (Industry)
Responsible Party: Sponsor
Other Study IDs: KIY-REG-001
Record Dates: First submitted 2018-06-10; First posted 2018-06-19 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cancer; Ovarian Cancer; Glioblastoma Multiforme; Anaplastic Astrocytoma
MeSH Terms: conditions — Ovarian Neoplasms; Glioblastoma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Fresh tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor tissue tested with EV3D Assay: Cancer tissue from multiple sites in the body, to include ovarian, brain, and other rare tumors.
  Interventions: Diagnostic Test: EV3D Assay

INTERVENTIONS:
Diagnostic Test: EV3D Assay — The EV3D assay uses freshly obtained tumor specimen to predict tissue drug response.

SUMMARY:
This is a prospective, non-randomized, observational registry study evaluating a patient-specific ex vivo 3D (EV3D) assay for drug response using a patient's own biopsy or resected tumor tissue for assessing tissue response to therapy in patients with advanced cancers, including ovarian cancer, high-grade gliomas, and high-grade rare tumors.

DETAILED DESCRIPTION:
This protocol defines a prospective, open-label, multi-institutional, non-interventional study for the purpose of examining the Assay's clinical use and potential to impact patient outcomes. This Study will establish a registry of clinical parameters, including clinical response, clinical outcomes, Assay performance and potential utilization across multiple types of advanced cancers in consenting patients who have their tumor tissue tested by the Assay. Physicians may have access to Assay results which which predict therapeutic response to cancer drugs most often prescribed to treat the specified indications. For cancers with standard of care (SOC) cancer drug treatments, the Assay panel tests SOC systemic agents per NCCN guidelines, some of which may include both FDA approved and off-label FDA approved therapies. The Assay currently assesses the most common cancer drugs across multiple tumor types. It requires freshly obtained tumor specimen that has not been previously preserved for traditional histologic analysis. The Registry will focus initially on tumor types and agents which have been analytically validated with the Assay and determined to meet strict laboratory qualifications and standards. The Registry will collect data on a limited number of cancer types to include epithelial ovarian cancer (EOC), high-grade gliomas (HGG) limited to anaplastic astrocytoma (AA) and glioblastoma multiforme (GBM), and high-grade rare tumors (RT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of or suspected diagnosis of EOC, HGG, high-grade RT
* Individual must undergo elective surgery or biopsy to remove tumor tissue
* Consideration as a candidate for systemic therapy with cytotoxic chemotherapy, targeted small molecule inhibitors or immunotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 3
* Written informed consent in accordance with institutional standards must be obtained from the patient or legal guardian

Exclusion Criteria:

* Inability or refusal of the patient or legal guardian to sign a written informed consent
* Failure to have surgery or a biopsy as part of routine clinical practice
* Refusal to have the Assay performed on their tissue
* Known active cancer metastatic to the brain except for patients with brain metastases that have been treated and are considered stable.
* Inability or unwillingness to receive chemotherapy treatment beyond surgery
* Any coincidental medical condition that, in the Investigator's opinion, would preclude participation in the study or compromise the patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected, newly diagnosed or relapsed diagnosis of advanced cancer (ovarian, brain, or other rare tumors) undergoing surgery or biopsy to remove tumor tissue will be enrolled and their tissue collected and tested with the EV3D Assay across drugs that are most often used to treat the specified cancer types, including standard of care therapies or as recommended by NCCN guidelines.
Sampling Method: Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Establish correlation of Assay results with patient outcomes | 2 year
  Compare Assay results to reported patient outcomes

SECONDARY OUTCOMES:
Evaluate the use of Assay results and the effects on medical decision-making and patient outcomes | 2 year
  Determine potential effect of Assay results on treatment plan
Compare clinical response (progression free survival or time to progression) in patients who receive treatment aligned with Assay results of response versus patients who are not treated aligned with Assay results of response | 2 years
  Compare Assay results to study patient clinical response
Compare clinical response (progression free survival or time to progression) in patients who receive treatment aligned with Assay results of response versus historical response rates | 2 years
  Compare Assay results to historical clinical response rates
Compare clinical outcomes (event free survival and overall survival) in patients who are treated aligned with Assay results versus historical response rates | 2 years
  Compare survival of study patients aligned with Assay results to historical survival rates
Define Assay success across histologic subtypes and classes of anti-cancer compounds | 2 years
  Evaluate Assay success rate

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Arkansas for Medical Sciences, Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Capital Health Institute for Neurosciences, Trenton, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Oregon Health & Science University, Portland, Oregon
  - Veterans Administration Portland Health Care System, Portland, Oregon
  - Penn State Health, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shuford S, Wilhelm C, Rayner M, Elrod A, Millard M, Mattingly C, Lotstein A, Smith AM, Guo QJ, O'Donnell L, Elder J, Puls L, Weroha SJ, Hou X, Zanfagnin V, Nick A, Stany MP, Maxwell GL, Conrads T, Sood AK, Orr D, Holmes LM, Gevaert M, Crosswell HE, DesRochers TM. Prospective Validation of an Ex Vivo, Patient-Derived 3D Spheroid Model for Response Predictions in Newly Diagnosed Ovarian Cancer. Sci Rep. 2019 Aug 1;9(1):11153. doi: 10.1038/s41598-019-47578-7. PMID 31371750
- [Result] Shuford S, Lipinski L, Abad A, Smith AM, Rayner M, O'Donnell L, Stuart J, Mechtler LL, Fabiano AJ, Edenfield J, Kanos C, Gardner S, Hodge P, Lynn M, Butowski NA, Han SJ, Redjal N, Crosswell HE, Vibat CRT, Holmes L, Gevaert M, Fenstermaker RA, DesRochers TM. Prospective prediction of clinical drug response in high-grade gliomas using an ex vivo 3D cell culture assay. Neurooncol Adv. 2021 May 7;3(1):vdab065. doi: 10.1093/noajnl/vdab065. eCollection 2021 Jan-Dec. PMID 34142085
- [Result] Reed MR, Lyle AG, De Loose A, Maddukuri L, Learned K, Beale HC, Kephart ET, Cheney A, van den Bout A, Lee MP, Hundley KN, Smith AM, DesRochers TM, Vibat CRT, Gokden M, Salama S, Wardell CP, Eoff RL, Vaske OM, Rodriguez A. A Functional Precision Medicine Pipeline Combines Comparative Transcriptomics and Tumor Organoid Modeling to Identify Bespoke Treatment Strategies for Glioblastoma. Cells. 2021 Dec 2;10(12):3400. doi: 10.3390/cells10123400. PMID 34943910
- See also: Prospective Validation of an Ex Vivo, Patient-Derived 3D Spheroid Model for Response Predictions in Newly Diagnosed Ovarian Cancer — https://www.nature.com/articles/s41598-019-47578-7
- See also: Prospective prediction of clinical drug response in high-grade gliomas using an ex vivo 3D cell culture assay — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8207705/pdf/vdab065.pdf